CLINICAL TRIAL: NCT03644810
Title: The Efficiency of Conditioned Pain Modulation is Associated With Levels of Pain Catastrophizing in Patients With Chronic Low Back Pain
Brief Title: The Association Between Conditioned Pain Modulation and Pain Catastrophizing in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Spine Centre of Southern Denmark (Other)
Responsible Party: Principal Investigator, Thorvaldur Skuli Palsson, Principal Investigator, Aalborg University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S-20170021
Record Dates: First submitted 2018-08-14; First posted 2018-08-23 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Catastrophizing Pain; Pain, Somatic; Chronic Low Back Pain
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Intervention Model Description: The study has a cross-sectional design and includes individuals (males and females) with and without chronic low back pain into two, equally large groups
Who Masked: Participant
Masking Description: The participants are blind to the study hypothesis and therefore the expected outcome of the tests performed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic low back pain (Active Comparator): Individuals with chronic low back pain. Baseline assessment of pain intensity, function, pain duration and pain catastrophizing thoughts is performed
  Pain sensitivity at the back and lower leg is measured at baseline and immediately after performing the cold pressor test
  Interventions: Diagnostic Test: PPT measurement; Diagnostic Test: Pain catastrophizing scale; Procedure: Cold Pressor Test
- Healthy controls (Active Comparator): Healthy, pain-free individuals who are age and gender matched to the low back pain group fill out the pain catastrophizing scale
  Pain sensitivity at the back and lower leg is measured at baseline and immediately after performing the cold pressor test
  Interventions: Diagnostic Test: PPT measurement; Diagnostic Test: Pain catastrophizing scale; Procedure: Cold Pressor Test

INTERVENTIONS:
Diagnostic Test: PPT measurement — The sensitivity to pressure which is gradually increased is assessed. The procedure is performed at the back and the lower leg
  Other Names: Assessment of pain sensitivity
Diagnostic Test: Pain catastrophizing scale — A validated questionnaire that measures three domains of pain-related catastrophizing thoughts: helplessness, rumination and excessive magnification
Procedure: Cold Pressor Test — The participant submerges one hand into a tank of cold (5 deg C), circulating water. The procedure is commonly know to decrease the sensitivity to pressure (PPT procedure) so that a difference appears in pain sensitivity when comparing PPT values before and after the procedure

SUMMARY:
This study evaluates the potential association between pain catastrophizing thoughts and the ability to dampen pain via endogenous descending inhibition. Half of the participants are persons with chronic low back pain and the other half are age and gender-matched controls

DETAILED DESCRIPTION:
Pain catastrophizing is a cognitive feature commonly seen in various musculoskeletal pain population and is considered an important factor to account for in rehabilitation. The ability to dampen pain via endogenous pain modulatory mechanisms is likewise known to be reduced in musculoskeletal pain conditions.

Studies utilizing functional magnetic resonance imaging (fMRI) have demonstrated that the supraspinal areas involved in pain-related cognitive processing to a great extent overlap with those involved in endogenous pain modulation. Therefore, it is plausible that factors such as pain catastrophizing thoughts may affect the nervous systems ability to dampen pain.

Chronic low back pain is the single clinical problem with the biggest impact in the modern society. Previous studies have demonstrated that pain catastrophizing and reduced endogenous pain inhibition are part of the clinical picture. However, previous studies have never investigated a potential relationship between these two factors.

ELIGIBILITY:
Inclusion Criteria:

Low back pain group:

* chronic low back pain ( lasting more than 3 months)
* intensity of ≥ 3/10 on a numeric rating scale
* pain is located in the area between the gluteal folds below to the thoracolumbal junction above.

Controls:

No current or previous history of musculoskeletal pain of ongoing nature

Exclusion Criteria:

Applies for both groups:

* Signs of radicular pain or other specific medical conditions e.g. rheumatologic disease or diabetes
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Association between levels of pain catastrophizing thoughts and endogenous pain inhibition | One session (45 min)
  The pain catastrophizing scale score is correlated with the changes in Pressure Pain Thresholds before and after the cold pressor test
  See descriptions of each assessment method below (outcome 2 and outcome 3, respectively)

SECONDARY OUTCOMES:
Changes in pressure pain thresholds (determined with pressure algometry) before and after the cold pressor test | 30 minutes
  Pressure Pain Thresholds (PPT) are assessed before and after the cold pressor test
  PPT measure the pressure needed to experience the first instance of pain. For this purpose, a pressure algometer (a pistol-like device with a 1cm2 contact surface) is used. Higher levels of pressure reflect lower pain sensitivity.
  In the cold pressor test, the subject is asked to submerge one hand into circulating water (constant temperature: 4 degrees C) for 2 minutes. When removing it from the water, the subject is asked to indicate the perceived pain using a numeric rating scale (see below). Before and after the cold pressor test, the PPT measurements are performed. The difference in PPT values before and after the cold pressor test is used in the correlation analysis described in outcome 1.
  The numeric rating scale is used to determine the perceived pain intensity from the cold water. The scale is runs from 0 - 10 where 0 is anchored with no pain and 10 reflects the worst pain imaginable
Catastrophizing thoughts measured with the Pain Catastrophizing Scale | 15 minutes
  The pain catastrophizing score by filling out the pain catastrophizing scale.The pain catastrophizing scale consists of 13 sentences describing pain-related thoughts or feelings. These are divided into 3 domains: rumination, magnification and helplessness. The subject is asked to indicate how how well each sentence applies for them: 0 = not at all, 1 = to a slight degree, 2 = to a moderate degree, 3 = to a great degree and 4 = all the time.
  The total score on the questionnaire can lie between 0 - 52 where a higher score indicates higher levels of pain catastrophizing thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Thorvaldur S Palsson, PhD, Principal Investigator — Aalborg University
Locations (1):
- Spine Centre of Southern Denmark, Middelfart, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
There are currently no plans on sharing data from this study with other researchers

REFERENCES:
- [Background] Edwards RR, Smith MT, Stonerock G, Haythornthwaite JA. Pain-related catastrophizing in healthy women is associated with greater temporal summation of and reduced habituation to thermal pain. Clin J Pain. 2006 Oct;22(8):730-7. doi: 10.1097/01.ajp.0000210914.72794.bc. PMID 16988570
- [Result] Vaegter HB, Palsson TS, Graven-Nielsen T. Facilitated Pronociceptive Pain Mechanisms in Radiating Back Pain Compared With Localized Back Pain. J Pain. 2017 Aug;18(8):973-983. doi: 10.1016/j.jpain.2017.03.002. Epub 2017 Mar 24. PMID 28344100
- [Result] Meints SM, Wang V, Edwards RR. Sex and Race Differences in Pain Sensitization among Patients with Chronic Low Back Pain. J Pain. 2018 Dec;19(12):1461-1470. doi: 10.1016/j.jpain.2018.07.001. Epub 2018 Jul 17. PMID 30025944
- [Result] Mlekusch S, Neziri AY, Limacher A, Juni P, Arendt-Nielsen L, Curatolo M. Conditioned Pain Modulation in Patients With Acute and Chronic Low Back Pain. Clin J Pain. 2016 Feb;32(2):116-21. doi: 10.1097/AJP.0000000000000238. PMID 26741741
- [Result] Correa JB, Costa LO, de Oliveira NT, Sluka KA, Liebano RE. Central sensitization and changes in conditioned pain modulation in people with chronic nonspecific low back pain: a case-control study. Exp Brain Res. 2015 Aug;233(8):2391-9. doi: 10.1007/s00221-015-4309-6. Epub 2015 May 12. PMID 25963754